CLINICAL TRIAL: NCT01477034
Title: Vitamin D and Adipose Tissue Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Kratz, Mario, Assistant Member, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UW NORC P&F KRATZ; 7598 (Other: FHCRC)
Record Dates: First submitted 2011-11-01; First posted 2011-11-22 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Vitamin D Deficiency; Obesity; Type 2 Diabetes Mellitus; Intestinal Permeability
Keywords: Vitamin D deficiency; Obesity; Inflammation; Low-grade, chronic inflammation; Adipose tissue inflammation; Diabetes; Type 2 diabetes mellitus; Insulin resistance; Intestinal permeability
MeSH Terms: conditions — Vitamin D Deficiency; Obesity; Diabetes Mellitus, Type 2; Inflammation; Diabetes Mellitus; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2,000 IU/day vitamin D3 x 6 months (Experimental): Subjects will take a 2,000 IU daily vitamin D3 supplement for 6 months.
  Interventions: Dietary Supplement: Vitamin D3
- 4,000 IU/day vitamin D3 x 6 months (Experimental): Subjects will take a 4,000 IU daily vitamin D3 supplement for 6 months.
  Interventions: Dietary Supplement: Vitamin D3
- 2,000 IU/day vitamin D3 x 3 months (Experimental): Subjects will take a 2,000 IU daily vitamin D3 supplement for 3 months.
  Interventions: Dietary Supplement: Vitamin D3
- 4,000 IU/day vitamin D3 x 3 months (Experimental): Subjects will take a 4,000 IU daily vitamin D3 supplement for 3 months.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 2,000 or 4,000 IU/day vitamin D3 for 3 or 6 months.
  Other Names: Carlson Labs Vitamin D3 capsules (2,000/4,000 IU/capsule)

SUMMARY:
Chronic, low-grade adipose tissue inflammation is a major risk factor for type 2 diabetes mellitus. The cause of adipose tissue inflammation has remained largely unclear. We hypothesize that vitamin D deficiency predisposes individuals to the development of adipose tissue inflammation, and that treatment of vitamin D deficient subjects with high dose vitamin D will reduce adipose tissue inflammation.

DETAILED DESCRIPTION:
The objective of this project is to investigate whether vitamin D modulates chronic low-grade adipose tissue inflammation in overweight and obese, vitamin D deficient men and women.

Obesity is associated with insulin resistance and an increased risk for type 2 diabetes mellitus. Numerous studies, mostly conducted in mouse models of obesity, strongly suggest that chronic low-grade inflammation of adipose and other tissues is the major mechanism by which increased adiposity is linked to insulin resistance. Adipose tissue inflammation may therefore be a promising therapeutic target to reduce insulin resistance and the risk of type 2 diabetes mellitus in obese individuals.

Based on several lines of evidence, we hypothesize that vitamin D is an environmental factor that affects the course of the inflammatory response in most tissues of the body, including adipose tissue. In our previous studies, we found that circulating plasma concentrations of 25-hydroxy vitamin D (25-OH-D) and the primary degradation product 24,25-dihydroxy vitamin D (24,25-OH2-D) were significantly associated with adipose tissue expression of adiponectin and negatively with TNF-alpha, even when adjusted for body mass index. Because these previous studies were cross-sectional, it is critical to complete an intervention study in humans to determine whether the observed association of vitamin D levels and adipose tissue inflammation is causal. The objectives of this pilot study are therefore to collect relevant preliminary data, and to begin an exploration of the mechanisms underlying this association such as intestinal permeability.

Increased intestinal permeability may contribute to chronic low-grade inflammation and signaling through the vitamin D receptor plays an important role in the maintenance of intestinal integrity. We will assess whether normalization of vitamin D status is associated with changes in intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years;
* BMI ≥25 kg/m2;
* Plasma 25-OH-vitamin D between 7 and 20 ng/mL
* Weight stable to within 10 pounds for 6 months prior to entering the study, and within 30 pounds of their lifetime maximum weight (excluding pregnancy);
* Ability to be admitted for ~6.5 hours on three occasions to the FHCRC Prevention Center,
* Ability to provide informed written consent;
* Willingness to take vitamin D3 capsules daily for 6 months

Exclusion Criteria:

* Chronic disease such as thyroid disease, liver disease, or kidney disease;
* Diabetes mellitus, or fasting glucose >125 mg/dL;
* Chronic inflammatory condition such as autoimmune disease or inflammatory bowel disease;
* Malabsorption syndromes (untreated celiac disease; condition after stomach or intestinal resection);
* Current or recent (within one month) chronic intake of medications likely to interfere with study endpoints [(insulin, antidiabetics, anabolic steroids, glucocorticosteroids, statins, blood thinners (warfarin, aspirin), non-steroidal anti-inflammatory drugs (if daily)];
* Current or recent (within 3 months) intake of vitamin D in excess of 600 IU/day;
* Anemia, recent history (within 3 months) of anemia; recent (within 3 months) blood donation; recent (within 3 months) participation in another study that involved blood draws; or plans to participate in other research that involves blood draws during the study period;
* Pregnancy in the last 6 months, plans to become pregnant during the study period, or current breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Tumor Necrosis Factor alpha expression in adipose tissue | Change from baseline to the 6 month visit
  Total RNA will be extracted from whole adipose tissue. TNF alpha mRNA will be quantified using PCR, and normalized using a normalization factor based on three housekeeping genes. We will compute the change in adipose tissue TNF alpha mRNA level between baseline and the 6 month visit.
Tumor Necrosis Factor alpha expression in adipose tissue | Change from baseline to the 3 month visit
  Total RNA will be extracted from whole adipose tissue. TNF alpha mRNA will be quantified using PCR, and normalized using a normalization factor based on three housekeeping genes. We will compute the change in adipose tissue TNF alpha mRNA level between baseline and the 3 month visit.

SECONDARY OUTCOMES:
Plasma concentrations of 24,25-dihydroxy vitamin D [24,25(OH)2D] | Change from baseline to the 6 month visit
  The concentration of 24,25(OH)2D will be measured in fasting plasma using high performance liquid chromatography-tandem mass spectometry (LC/MS/MS).
Adipose tissue concentration of 25-hydroxy vitamin D [25(OH)D] | Change from baseline to the 6 month visit
  Adipose tissue 25(OH)D will be measured using high performance liquid chromatography-tandem mass spectometry (LC/MS/MS.)
CD16+ macrophages in adipose tissue | Change from baseline to the 6 month visit
  The number or CD16+ macrophages in adipose tissue, normalized to the total number of CD14+CD206+ macrophages or the total number of CD45+ cells, will be measured using multi-parameter flow cytometry.
CD8+ T cells in adipose tissue | Change from baseline to the 6 month visit
  The number of CD8+ T cells in adipose tissue, normalized to the total number of CD3+ cells, will be measured using multi-parameter flow cytometry.
Plasma concentration of 25-hydroxy vitamin D [25(OH)D] | Change from baseline to the 6 month visit
  Plasma 25(OH)D will be measured by high performance liquid chromatography-tandem mass spectometry (LC/MS/MS).
Adipose tissue concentration of cholecalciferol (vitamin D3) | Change from baseline to the 6 month visit
  Adipose tissue concentrations of cholecalciferol will be measured by high performance liquid chromatography-tandem mass spectometry (LC/MS/MS)
CD11c+ macrophages in adipose tissue | Change from baseline to the 6 month visit
  The number of CD11c+ macrophages in adipose tissue, normalized to the total number of CD45+ cells, will be measured by multi-parameter flow cytometry.
CD4+CD25+ T cells in adipose tissue | Change from baseline to the 6 month visit
  The number of CD4+CD25+ T cells in adipose tissue, normalized to the total number of CD4+ T cells, will be measured by multi-parameter flow cytometry.
Intestinal permeability, as assessed by the 5-hour urinary lactulose/mannitol test | Change from baseline to 6 month clinic visit.
  Intestinal permeability will be assessed at each clinic visit by administering 2g of mannitol and 5 g of lactulose to the oral glucose tolerance test beverage followed by collection of urine for 5 hours afterwards. Recovery of mannitol and lactulose in urine will be measured by gas chromatography, and will be indicative of the degree of intestinal permeability.
Fasting plasma zonulin concentrations | Change from baseline to 6 month clinic visit
  Zonulin concentrations will be measured by enzyme-linked immunosorbent assay in fasting plasma collected at all clinic visits. Plasma zonulin is a marker of intestinal permeability.
Fasting plasma lipopolysaccharide binding protein (LBP) | Change from baseline to 6 month clinic visit
  Lipopolysaccharide binding protein (LBP) will be measured by enzyme-linked immunosorbent assay in fasting plasma collected at all clinic visits. LBP is an acute phase protein secreted by the liver in response to endotoxin (lipopolysaccharide) exposure.
Plasma concentrations of 24,25-dihydroxy vitamin D [24,25(OH)2D] | Change from baseline to the 3 month visit
  The concentration of 24,25(OH)2D will be measured in fasting plasma using high performance liquid chromatography-tandem mass spectometry (LC/MS/MS).
Adipose tissue concentration of 25-hydroxy vitamin D [25(OH)D] | Change from baseline to the 3 month visit
  Adipose tissue 25(OH)D will be measured using high performance liquid chromatography-tandem mass spectometry (LC/MS/MS.)
CD16+ macrophages in adipose tissue | Change from baseline to the 3 month visit
  The number or CD16+ macrophages in adipose tissue, normalized to the total number of CD14+CD206+ macrophages or the total number of CD45+ cells, will be measured using multi-parameter flow cytometry.
CD8+ T cells in adipose tissue | Change from baseline to the 3 month visit
  The number of CD8+ T cells in adipose tissue, normalized to the total number of CD3+ cells, will be measured using multi-parameter flow cytometry.
Plasma concentration of 25-hydroxy vitamin D [25(OH)D] | Change from baseline to the 3 month visit
  Plasma 25(OH)D will be measured by high performance liquid chromatography-tandem mass spectometry (LC/MS/MS).
Adipose tissue concentration of cholecalciferol (vitamin D3) | Change from baseline to the 3 month visit
  Adipose tissue concentrations of cholecalciferol will be measured by high performance liquid chromatography-tandem mass spectometry (LC/MS/MS)
CD11c+ macrophages in adipose tissue | Change from baseline to the 3 month visit
  The number of CD11c+ macrophages in adipose tissue, normalized to the total number of CD45+ cells, will be measured by multi-parameter flow cytometry.
CD4+CD25+ T cells in adipose tissue | Change from baseline to the 3 month visit
  The number of CD4+CD25+ T cells in adipose tissue, normalized to the total number of CD4+ T cells, will be measured by multi-parameter flow cytometry.
Intestinal permeability, as assessed by the 5-hour urinary lactulose/mannitol test | Change from baseline to 3 month clinic visit.
  Intestinal permeability will be assessed at each clinic visit by administering 2g of mannitol and 5 g of lactulose to the oral glucose tolerance test beverage followed by collection of urine for 5 hours afterwards. Recovery of mannitol and lactulose in urine will be measured by gas chromatography, and will be indicative of the degree of intestinal permeability.
Fasting plasma zonulin concentrations | Change from baseline to 3 month clinic visit
  Zonulin concentrations will be measured by enzyme-linked immunosorbent assay in fasting plasma collected at all clinic visits. Plasma zonulin is a marker of intestinal permeability.
Fasting plasma lipopolysaccharide binding protein (LBP) | Change from baseline to 3 month clinic visit
  Lipopolysaccharide binding protein (LBP) will be measured by enzyme-linked immunosorbent assay in fasting plasma collected at all clinic visits. LBP is an acute phase protein secreted by the liver in response to endotoxin (lipopolysaccharide) exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kratz, Ph.D., Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Best CM, Riley DV, Laha TJ, Pflaum H, Zelnick LR, Hsu S, Thummel KE, Foster-Schubert KE, Kuzma JN, Cromer G, Larson I, Hagman DK, Heshelman K, Kratz M, de Boer IH, Hoofnagle AN. Vitamin D in human serum and adipose tissue after supplementation. Am J Clin Nutr. 2021 Jan 4;113(1):83-91. doi: 10.1093/ajcn/nqaa295. PMID 33184642